CLINICAL TRIAL: NCT05661890
Title: Prevalence of Seasonal Influenza and Pneumococcal Vaccination and Determinants of Vaccination in the Elderly: Nested Case-Control Study
Brief Title: Seasonal Influenza and Pneumococcal Vaccination in the Elderly
Status: Completed | Type: Observational
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Belgin Akın, Professor, Lokman Hekim University
Other Study IDs: LokmanHekimU-SBF-HB-BA-01
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Immunization; Infection; Influenza; Pneumonia; Vaccine Refusal
Keywords: Vaccine; Influenza; Pneumonia; Elderly
MeSH Terms: conditions — Infections; Influenza, Human; Pneumonia; Vaccination Refusal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The elderly population and individuals with chronic diseases are at high risk for influenza and influenza-related pneumonia, and it is emphasized that taking pneumonia and influenza vaccine together is effective in reducing mortality as well as hospitalization rates and costs due to pneumonia, influenza, and congestive heart disease.

This study that will be carried out will enable to determine the population-based prevalence of the relevant vaccines in the elderly and to determine the determinants of vaccination with the case group to be determined based on this.

The aim of the study is two phases.

1. Determination of the prevalence of seasonal influenza and pneumococcal vaccination in elderly people over the over the age of 65 living in Ankara.
2. Investigation of socioeconomic characteristics and vaccine indecision and some health-related determinants of vaccination through the case group created based on the preliminary study on the prevalence of seasonal influenza and pneumococcal vaccination in the elderly over the age of 65 living in Ankara.

The study, which includes cross-sectional prevalence and retrospective case-control stages, is planned to be carried out with individuals over the age of 65 living in Ankara province between November 1 and December 31, 2022.

DETAILED DESCRIPTION:
The elderly population and individuals with chronic diseases are at high risk for influenza and influenza-related pneumonia, and it is emphasized that taking pneumonia and influenza vaccine together is effective in reducing mortality as well as hospitalization rates and costs due to pneumonia, influenza, and congestive heart disease.

In recent years, progress has been made in vaccination as a result of the increase in health-seeking behavior due to the pandemic, the greater importance of influenza and pneumococcal vaccine application recommendations, and the perception of the prevention of lung infections due to COVID-19.

However, the discussions on the need to predict vaccine demand and examine health behaviors, health education, and research on new methods of vaccination efficacy in reducing future epidemics continue to be relevant.

This study that will be carried out will enable to determine the population-based prevalence of the relevant vaccines in the elderly and to determine the determinants of vaccination with the case group to be determined based on this.

Research questions-Prevalence

1. What is the prevalence of influenza vaccination in the elderly?
2. What is the prevalence of pneumonia vaccination in the elderly?

Research Questions - Case Control

1. Are socio-economic characteristics (region of residence, monthly income, education, perceived economic status) effective in vaccinating the elderly?
2. Are health-related features (chronic illness, drug use, previous vaccination status, priority preference in health care, frequency of hospitalization and hospitalization in the last six months, distance from health institution, self-defense behavior) effective in vaccinating the elderly?
3. Is the vaccination attitude effective in vaccinating the elderly?

ELIGIBILITY:
Inclusion Criteria:

-Over the age of 65.

Exclusion Criteria:

* Cancer diagnosis
* Having a disease that will require immunosuppressive treatment
* Transplantation cases
* Rheumatoid arthritis
* Systemic lupus erythematosus
* Inflammatory bowel disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The population is individuals over the age of 65 living in the central district of Ankara.
  The sample size required for the study and its distribution by neighborhoods were calculated according to the WHO LKT modüle. The minimum required sample size was calculated as 972, by accepting the preliminary decision that 75 lots would be used in the study, and p=35%, 95% confidence interval, and deviation value of ±3 in the study. However, the minimum sample size for the number of elderly per LOT was accepted as 15 and the number was increased by 20% considering possible data losses and the sample size was accepted as 1166.
  The region of each lot was determined on the map, and sample selection was made using random methods in the study.
Sampling Method: Probability Sample
Enrollment: 1166 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Number of Influenza Vaccination uptake | During 2022
  The number of self reported influenza vaccine uptake

CONTACTS AND LOCATIONS:
Overall Officials: Belgin Akın, Principal Investigator — Lokman Hekim University
Locations (1):
- Lokman Hekim University, Ankara, Çankaya, Turkey (Türkiye)